CLINICAL TRIAL: NCT00691730
Title: The Role of VEGF-A Signaling in Maintenance of the Glomerular Filtration Barrier and Blood Pressure
Brief Title: Kidney and Blood Pressure Changes in Patients Receiving Bevacizumab, Aflibercept, Sunitinib, or Cediranib for Cancer
Acronym: NCI 8076
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PHL-064; NCI-2009-00277 (Other: CTRP (Clinical Trials Reporting System)); PMH-PHL-064; CDR0000588665 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: laboratory biomarker analysis — Only sample collection, no other intervention - Correlative studies

SUMMARY:
This research study is looking at kidney and blood pressure changes in patients receiving bevacizumab, aflibercept, sunitinib, or cediranib for cancer. Studying samples of blood and urine from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment with an antiangiogenic drug.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To study the renal and blood pressure changes in patients treated with bevacizumab, aflibercept, sunitinib malate, or cediranib for their cancer.

II. To determine the physiological mechanisms behind proteinuria and hypertension induced by antiangiogenic therapies (i.e., rarefaction; imbalance in eNOS, prostacyclin [PGI_2], prostaglandin E2 [PGE_2], and thromboxane A2 [TXA2]; renin/aldosterone; or renovascular hypertension).

III. To determine whether soluble factors (like tyrosine kinase 1 [sFlt1], bFGF, and VEGF) and steady state drug concentration are predictive of the development of proteinuria/hypertension.

OUTLINE: This is a multicenter study.

Patients undergo blood and urine sample collection periodically. Urine samples are assessed for PGI2 and TXA2 levels using validated ELISA methods. Urine is also assessed for protein and creatinine levels, microalbumin, osmolality, and electrolytes. Blood samples are assessed for pharmacokinetics and sFlt1, VEGF, and bFGF levels by validated ELISA methods. Blood samples are also assessed for steady state drug concentration, renin, and aldosterone levels.

ELIGIBILITY:
Inclusion Criteria:

* Planning to start treatment with one of the following antiangiogenic drugs as single agents or in combination with chemotherapy for their cancer:

  * Cediranib (AZD2171 )
  * Bevacizumab (Avastin)
  * Sunitinib (Sutent)
  * Aflibercept (VEGF Trap)
* Urinalysis negative for protein OR 24-hour urine for protein < 500 mg
* Prior chemotherapy within the past 12 months allowed
* More than 12 months since prior antiangiogenic drugs, including monoclonal antibodies that bind to VEGF or tyrosine kinase inhibitors that block VEGFR2
* At least 6 weeks since prior and no concurrent aldosterone receptor antagonists (e.g., spironolactone [aldactone] or eplerenone)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are going to start treatment with bevacizumab, VEGF Trap, sunitinib or AZD2171.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Renal and blood pressure changes | Up to 8 weeks
Physiological mechanism behind proteinuria and hypertension induced by antiangiogenic therapies | Up to 8 weeks
Predictive value of soluble factors in the development of proteinuria or hypertension | Up to 8 weeks
Predictive value of steady state drug concentrations in the development of proteinuria or hypertension | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Moore, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (4):
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - London Regional Cancer Program, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario